CLINICAL TRIAL: NCT06503315
Title: Genetic Polymorphism in Matrix Metalloproteinase 9 in Chronic Obstructive Pulmonary Disease in Sohag University Hospital.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yassmin Ismail, demonastrator at department of biochemistry ,sohag university, Sohag University
Other Study IDs: Soh-Med-24-06-09MS
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: Clinical assessment is based on the presence of symptoms (low vs. high) and the previous history of exacerbation( ECOPD) (≤ 1 moderate ECOPD in the previous year vs. more than one severe (hospitalized) ECOPD). Using these two dimensions, GOLD 2023 proposes to classify COPD patients in one of three groups (A, B, or E) .
- control group: The control group includes 70 asymptomatic smokers and will be matched with cases by sex, age, smoking status, lacking chronic diseases in the respiratory system as malignancy and bronchial asthma

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a heterogeneous and complex disease with multiple clinical presentations or phenotypes and remains a highly prevalent condition, causing significant morbidity and mortality worldwide.

Chronic obstructive pulmonary disease (COPD) is the third most common cause of global mortality, affecting over 210 million individuals.

Chronic obstructive pulmonary disease (COPD) is a chronic airway disease involving chronic local and systemic inflammatory changes, clinically characterized by continuous and progressive airflow obstruction with airway remodeling and lung parenchyma destruction as pathological basis.

The precise molecular mechanism underlying the pathogenesis of COPD remains unclear ( Zhang J. et al., 2021). At present, it is generally believed that several risk factors are directly related to the pathogenesis of COPD, including host and environmental factors .

Among environmental factors, smoking, exposure to chemicals, indoor and outdoor air pollution are risk factors for COPD.

Host factors of COPD include antitrypsin-1, excessive deposition of extracellular matrix (ECM), corticosteroids, inflammatory stimuli, and metabolic imbalances .

Matrix metalloproteinases (MMPs) is a family of calcium- and zinc-dependent proteinase. There are currently at least 26 subtypes that can degrade almost all extracellular matrix and basement membrane components .

The MMP-9 gene is located on human chromosome 16, including 13 exons and 12 introns and its regulation mainly occurs at the transcriptional level. In the pathogenesis of COPD, MMP-9 mainly degrades the extracellular matrix and basement membrane of alveolar wall, destroying the normal structure of lung tissue. At the same time, MMP-9 also repairs the extracellular matrix and participates in respiratory tract reconstruction.

In addition, MMP-9 can also participate in inflammatory response, causing inflammatory cells to accumulate in the airway, thus increasing airway responsiveness. Study found that MMP-9 is highly expressed in the lung tissues of COPD patients and leads to generation of sputum. MMPs are important in COPD. They degrade matrix proteins (elastin, collagen) during the disease progression .

Therefore the analysis of MMP-9 gene polymorphism is an important starting point to explore the susceptibility to COPD. It has been found that there is a mutation from C to T at site 1562 of promoter MMP-9, which may affect the expression level of MMP-9 gene. The MMP-9-C1562T polymorphism is an important reason for the abnormal increase of MMP-9 expression level .

ELIGIBILITY:
Inclusion Criteria:

chronic respiratory symptom and signs such as cough ,breathlessness , wheeze ; forced expiratory volume in one second(FEV1)of predicted (FEV1%) less than 80 % ; the ratio of FEV1 to forced vital capacity (FVC , FEV1/ FVC)<70 % ; FEV1reversibility after inhalation of 200g salbutamol (bronchodilator) of less than 12 % of prebronchodilator FEV1.

Exclusion Criteria:

Coexistence of asthma and COPD or with earlier history of bronchial asthma as well as patients who have never smoked were excluded from the study.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: chronic respiratory symptom and signs such as cough ,breathlessness , wheeze ; forced expiratory volume in one second(FEV1)of predicted (FEV1%) less than 80 % ; the ratio of FEV1 to forced vital capacity (FVC , FEV1/ FVC)<70 % ; FEV1reversibility after inhalation of 200g salbutamol (bronchodilator) of less than 12 % of prebronchodilator FEV1.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Matrix metalloproteinase-9 gene polymorphism | 18 months
  Matrix metalloproteinase-9 gene polymorphism by conventional PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Agusti A, Bohm M, Celli B, Criner GJ, Garcia-Alvarez A, Martinez F, Sin DD, Vogelmeier CF. GOLD COPD DOCUMENT 2023: a brief update for practicing cardiologists. Clin Res Cardiol. 2024 Feb;113(2):195-204. doi: 10.1007/s00392-023-02217-0. Epub 2023 May 26. PMID 37233751
- [Background] Cabral-Pacheco GA, Garza-Veloz I, Castruita-De la Rosa C, Ramirez-Acuna JM, Perez-Romero BA, Guerrero-Rodriguez JF, Martinez-Avila N, Martinez-Fierro ML. The Roles of Matrix Metalloproteinases and Their Inhibitors in Human Diseases. Int J Mol Sci. 2020 Dec 20;21(24):9739. doi: 10.3390/ijms21249739. PMID 33419373
- [Background] Cai L, Zuo X, Ma L, Zhang Y, Xu F, Lu B. Associations of MMP9 polymorphism with the risk of severe pneumonia in a Southern Chinese children population. BMC Infect Dis. 2024 Jan 2;24(1):19. doi: 10.1186/s12879-023-08931-4. PMID 38166679
- [Background] Lu Z, Coll P, Maitre B, Epaud R, Lanone S. Air pollution as an early determinant of COPD. Eur Respir Rev. 2022 Aug 10;31(165):220059. doi: 10.1183/16000617.0059-2022. Print 2022 Sep 30. PMID 35948393